CLINICAL TRIAL: NCT05160064
Title: Long-term Longitudinal Cohort Registry of Patients Treated With Loncastuximab Tesirine
Brief Title: Long-term Registry of Patients Treated With Loncastuximab Tesirine
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor administrative decision
Sponsor: ADC Therapeutics S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: ADCT-402-N01
Record Dates: First submitted 2021-12-03; First posted 2021-12-16 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: B-Cell Lymphomas
Keywords: Diffuse Large B-Cell Lymphoma; Loncastuximab tesirine; Non-Hodgkin Lymphoma; Relapsed/Refractory Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 48 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients Treated with Loncastuximab Tesirine: Patients with B-cell lymphomas and other diagnoses who have been treated with loncastuximab tesirine will have their medical chart data entered into the registry.

SUMMARY:
Retrospective and prospective multi-center observational study of patients with B-cell lymphomas treated with loncastuximab tesirine treatment in real-world practice.

DETAILED DESCRIPTION:
The purpose of this study is to assess treatment patterns and generate evidence on the effectiveness and safety of loncastuximab tesirine treatment in real-world practice. This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Inclusion Criteria:

* Must be ≥ 18 years of age at the time of consent.
* Initiated or initiating commercially available loncastuximab tesirine treatment.
* Written informed consent must be obtained prior to any registry activities.

Exclusion Criteria:

* Prior loncastuximab tesirine exposure in clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients initiated or initiating commercially available loncastuximab tesirine treatment.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-06-30 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | Up to 48 Months
Overall Survival (OS) | Up to 48 Months
Duration of Response (DoR) | Up to 48 Months
Overall Response Rate (ORR) | Up to 48 Months
Time to Partial Response (PR) | Up to 48 Months
Time to Complete Response (CR) | Up to 48 Months
Time to Disease Progression | Up to 48 Months
Number of Patients with Adverse Events | Up to 48 Months
  Includes serious adverse events (SAEs) and adverse events (AEs) Grade 3 or higher for the events of: edema, myelosuppression, infections, and cutaneous reactions.

SECONDARY OUTCOMES:
Number of Hospitalizations | Up to 48 Months
Duration of Hospitalizations | Up to 48 Months
Reasons for Hospitalizations | Up to 48 Months
Number of Surgeries | Up to 48 Months
Type of Surgeries | Up to 48 Months
Reasons for Surgeries | Up to 48 Months
Number of Emergency Room Visits | Up to 48 Months
Reasons for Emergency Room Visits | Up to 48 Months
Number of Outpatient Visits | Up to 48 Months
Reasons for Outpatient Visits | Up to 48 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Compassionate Cancer Care Medical Group, Fountain Valley, California, United States

IPD SHARING:
Plan to Share IPD: No